CLINICAL TRIAL: NCT05955495
Title: Length of Stay Between Early Versus Delayed Oral Postoperative Feeding After Gynecologic Surgery Under General Anesthesia: Randomized Controlled Trial, Single Center
Brief Title: Length of Stay Between Early Versus Delayed Oral Postoperative Feeding
Acronym: LOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 002/2566
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Early Feeding
MeSH Terms: interventions — Food

STUDY DESIGN:
Intervention Model Description: The participants were randomized (1:1 computerized block randomization) into two groups. One group is early feeding and another is delayed feeding.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed feeding (Active Comparator)
  Interventions: Other: Food
- Early feeding (Experimental)
  Interventions: Other: Food

INTERVENTIONS:
Other: Food — Post-operative feeding includes water, liquid diet, soft diet.

SUMMARY:
Length of stay between early versus delayed oral postoperative feeding after gynecologic surgery under General Anesthesia: Randomized Controlled Trial, single center

The goal of this Randomized Controlled Trial is to compare Length of stay between early versus delayed oral postoperative feeding after gynecologic surgery under General Anesthesia. The main question[s] it aims to answer are:

* Length of stay
* Complications Participants will randomized (1:1 block randomization ) into Group A or B. The comparison groups are early and delayed postoperative feeding.

ELIGIBILITY:
Inclusion Criteria:

* Participants undergoing gynecologic surgery with stable vital signs
* Participants undergoing abdominal gynecologic surgery
* No evidence of malignancy
* No underlying disease relating to GI system
* Not currently having gut obstruction
* No previous abdominal surgeries aside from appendectomy
* Previous history of abdominal radiation

Exclusion Criteria:

* Transferred to ICU postoperatively
* on ETT, NG
* Participants with immediate complications from operation
* No informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women presenting with gynecologic condition.
Enrollment: 34 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Length of stay | 12 months
  Length of stay between early versus delayed oral postoperative feeding

SECONDARY OUTCOMES:
Complications | 12 months
  Complications occur during postoperative feeding between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Penpilai Vinitchaikul, MD, Principal Investigator — Queen SVMH
Locations (1):
- Chuenrutai Yeekian, Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Data were input in Excel spreadsheet and SPSS

REFERENCES:
- [Background] Charoenkwan K, Matovinovic E. Early versus delayed oral fluids and food for reducing complications after major abdominal gynaecologic surgery. Cochrane Database Syst Rev. 2014 Dec 12;2014(12):CD004508. doi: 10.1002/14651858.CD004508.pub4. PMID 25502897
- [Background] ACOG Committee Opinion No. 750: Perioperative Pathways: Enhanced Recovery After Surgery. Obstet Gynecol. 2018 Sep;132(3):e120-e130. doi: 10.1097/AOG.0000000000002818. PMID 30134426
- [Background] Chiewhatpong P, Charoenkwan K, Smithiseth K, Lapisatepun W, Lapisatepun P, Phimphilai M, Muangmool T, Cheewakriangkrai C, Suprasert P, Srisomboon J. Effectiveness of enhanced recovery after surgery protocol in open gynecologic oncology surgery: A randomized controlled trial. Int J Gynaecol Obstet. 2022 Nov;159(2):568-576. doi: 10.1002/ijgo.14211. Epub 2022 Apr 21. PMID 35396709
- [Background] Kehlet H, Wilmore DW. Evidence-based surgical care and the evolution of fast-track surgery. Ann Surg. 2008 Aug;248(2):189-98. doi: 10.1097/SLA.0b013e31817f2c1a. PMID 18650627
- [Background] Nelson G, Bakkum-Gamez J, Kalogera E, Glaser G, Altman A, Meyer LA, Taylor JS, Iniesta M, Lasala J, Mena G, Scott M, Gillis C, Elias K, Wijk L, Huang J, Nygren J, Ljungqvist O, Ramirez PT, Dowdy SC. Guidelines for perioperative care in gynecologic/oncology: Enhanced Recovery After Surgery (ERAS) Society recommendations-2019 update. Int J Gynecol Cancer. 2019 May;29(4):651-668. doi: 10.1136/ijgc-2019-000356. Epub 2019 Mar 15. PMID 30877144
- [Background] Hessov I, Rylev Larsen K, Sondergaard K. Improved early alimentation after radical hysterectomies without the traditional use of stomach tube. Acta Obstet Gynecol Scand. 1988;67(3):225-8. doi: 10.3109/00016348809004208. PMID 3140573
- [Background] Muallem MZ, Dimitrova D, Pietzner K, Richter R, Feldheiser A, Scharfe I, Schmeil I, Hosl TM, Mustea A, Wimberger P, Burges A, Kimmig R, Sehouli J. Implementation of Enhanced Recovery After Surgery (ERAS) Pathways in Gynecologic Oncology. A NOGGO-AGO* survey of 144 Gynecological Departments in Germany. Anticancer Res. 2016 Aug;36(8):4227-32. PMID 27466536
- [Background] Wijk L, Franzen K, Ljungqvist O, Nilsson K. Enhanced Recovery after Surgery Protocol in Abdominal Hysterectomies for Malignant versus Benign Disease. Gynecol Obstet Invest. 2016;81(5):461-7. doi: 10.1159/000443396. Epub 2016 Jan 23. PMID 26799328
- [Background] Kalogera E, Dowdy SC. Enhanced Recovery Pathway in Gynecologic Surgery: Improving Outcomes Through Evidence-Based Medicine. Obstet Gynecol Clin North Am. 2016 Sep;43(3):551-73. doi: 10.1016/j.ogc.2016.04.006. PMID 27521884
- [Background] Balayla J, Bujold E, Lapensee L, Mayrand MH, Sansregret A. Early Versus Delayed Postoperative Feeding After Major Gynaecological Surgery and its Effects on Clinical Outcomes, Patient Satisfaction, and Length of Stay: A Randomized Controlled Trial. J Obstet Gynaecol Can. 2015 Dec;37(12):1079-85. doi: 10.1016/s1701-2163(16)30073-1. PMID 26637080